CLINICAL TRIAL: NCT00712192
Title: The Impact on Endothelial Function and Integrity by Endoscopic Saphenous Vein Harvest for Coronary Artery Bypass Grafting
Brief Title: Endoscopic Saphenous Vein Harvest for Coronary Artery Bypass Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Shih-Hong Huang, Far Eastern Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 95016; FEMH - 95 - C -002
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2008-07

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery bypass grafting; endoscopic vein harvest; saphenous vein; endothelial cells; eNOS; ET-1
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: coronary artery bypass grafting — patient with coroary artery diseases underwent coronary artery bypass grafting surgery

SUMMARY:
Although the long saphenous vein remains the most commonly used conduit in coronary revascularization, traditional open vein harvest may lead to significantly impaired wound healing and post-operative pain. To this end, endoscopic saphenous vein harvesting techniques have been shown to reduce post-operative morbidity. Studies have shown that endothelial integrity and luminal nitric oxide synthase (NOS) are better preserved with novel "no-touch" techniques; however, the effect and the associated mechanism of endoscopic vein harvest on endothelial integrity and function remain unknown. Therefore, in the present proposal, we will collect the saphenous vein segements immediately after harvesting, reperfusion, and grafting, and then use enzyme-linked immunosorbant assay (ELISA), immunohistochemical staining (IHC), and real-time polymerase chain reaction (RT-PCR) to detect the expression and distribution of endothelial NOS (eNOS), endothelin-1 (ET-1), vascular cell adhesion molecule-1 (VCAM-1), intracellular adhesion molecule-1 (ICAM-1), and platelet endothelial cell adhesion molecule-1(PECAM-1) at protein and RNA levels in the endothelium of saphenous veins. The major aim of this study is to elucidate the effect and mechanism of endoscopic saphenous vein harvesting on endothelial properties as compare to conventional open vein harvest technique.

ELIGIBILITY:
Inclusion Criteria:

* patient with coronary artery disease underwent coronary artery bypass grafting in our hospital

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)